CLINICAL TRIAL: NCT01167491
Title: Activating Receptors and DAP12 Protein in Wegener's Granulomatosis
Brief Title: Study of One Protein Implicated in Wegener Disease
Acronym: DAP12WEGENER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: P081238
Record Dates: First submitted 2010-07-12; First posted 2010-07-22 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Wegener's Granulomatosis
Keywords: Wegener; CD4+ T cells; DAP12; NKG2D
MeSH Terms: conditions — Granulomatosis with Polyangiitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Disease group (Other): Physiopathology
  Interventions: Biological: Physiopathology Endpoint Classification

INTERVENTIONS:
Biological: Physiopathology Endpoint Classification — Blood samples will be collected during a routine medical visit.

SUMMARY:
The investigators recently showed an abnormal expansion of NK-like CD4+ T cells in Wegener's granulomatosis (WG), mainly in the diffuse vasculitis presentation. These cells expressed an assortment of activating NK cell receptors and their signaling partners, in particular DAP12. The investigators hypothesize that DAP12, or a downstream signaling target of DAP12, is the missing link between the different cell components involved in WG (neutrophils, macrophages, CD4 T cells).

DETAILED DESCRIPTION:
The investigators will test our hypothesis of "DAP-12 gain-of-function" by quantitative (mRNA and protein) and qualitative (DNA, signaling and cellular activation) analysis of the DAP12 signaling pathway in WG patients with localized (group 1; n=30) or diffuse WG (group 2; n=30) by comparison with patients with micro polyangitis (group 3; n=30), or with sarcoidosis ( group 4; n=30), and healthy blood donors (group 5; n=30). Blood samples will be collected during a routine medical visit. These results may help to design future therapeutic strategies based on modulation of specific intra-cellular pathways involved in the disease.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: WG, with granulomatous lesions limited to upper airway or lungs and no evidence of generalized vasculitis ,± biopsy, ± anti-PR3 ANCA
* Group 2: WG with granulomatous lesions plus vasculitis expression (renal, neurological, skin, gut or heart involvement), ± biopsy, ± anti-PR3 ANCA
* Group 3: Necrotizing vasculitis with no granulomatous lesions, ± PAUCI immune glomerulonephritis, ± anti-MPO ANCA
* Group 4: clinical presentation compatible with sarcoidosis, ± biopsy, ± ECA elevated ± tuberculin anergy

Exclusion Criteria:

* <18 years
* Pregnancy or breastfeeding
* Absence of signed informed consent
* No affiliation to insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2010-05; Primary Completion 2013-11 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
level of mRNA expression of DAP12 | less than 24 hours
  Measure:level of mRNA expression of DAP12 by RT-PCR in CD4+T cells, macrophages and neutrophils

SECONDARY OUTCOMES:
level of expression of DAP 12 downstream signalling proteins | Less than 24 hours
  Measure: level of expression of DAP 12 downstream signalling proteins in CD4+ T cells, macrophages and neutrophils

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde De Menthon,, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Medecine Interne Hôpital Saint Louis, Paris, France